CLINICAL TRIAL: NCT04077814
Title: Association Between the Transcranial Direct Current Stimulation (tDCS) and Foot Drop Stimulation (FDS) for Gait Rehabilitation After Stroke - A Randomized Clinical Trial
Brief Title: Association Between the tDCS and FDS for Gait Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Aline de Souza Pagnussat, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tDCS_FDS_2018
Record Dates: First submitted 2019-06-12; First posted 2019-09-04 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: Cerebrovascular Accident; Cerebrovascular Stroke; Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ShamtDCS+FDS (Active Comparator): Chronic stroke patients submitted to Foot Drop Stimulation (FDS) + Sham Transcranial direct brain stimulation (tDCS)
  Interventions: Device: Foot Drop Stimulatio - Neuro Orthosis
- tDCS+FDS (Experimental): Chronic stroke patients submitted to Foot Drop Stimulation (FDS) + Transcranial direct brain stimulation (tDCS)
  Interventions: Device: Foot Drop Stimulatio - Neuro Orthosis; Device: Transcranial direct brain stimulation

INTERVENTIONS:
Device: Foot Drop Stimulatio - Neuro Orthosis — Walkaide is the Foot drop stimulator (FDS) on the peroneal nerve provides active dorsiflexion of muscle during the swing phase of gait.
Device: Transcranial direct brain stimulation — Transcranial direct brain stimulation on motor cortex
  Arms: tDCS+FDS

SUMMARY:
The aim of this study is to verify the effectiveness of tDCS combined with foot drop stimulation (FDS) on gait rehabilitation of post-stroke subjects with mild and moderate compromise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ischemic or hemorrhagic stroke diagnosis.
* Mild, moderate or severe hemiparesis (chronic stroke - at least 6 months)
* Minimal cognitive ability to understand commands
* Able to walk 10 meters unassisted or with minimal assistance

Exclusion Criteria:

* No current use of antiepileptic drugs for seizures
* Secondary musculoskeletal disorder involving the lower limb
* Contraindication for electrical stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Kinematic gait anaysis. | The outcome will assess at baseline and two weeks after the intervention. One month later that finished the intensive treatment subjects will re-evaluate.
  Evaluated by means of the 3-D motion analysis system (BTS SMART DX 400)

SECONDARY OUTCOMES:
Kinetic gait anaysis. | The outcome will assess at baseline and two weeks after the intervention. One month later that finished the intensive treatment subjects will re-evaluate.
  Assessed by force platform (BTS P-6000)
Postural Control | The outcome will assess at baseline and two weeks after the intervention. One month later that finished the intensive treatment subjects will re-evaluate.
  Evaluated by Center of Pressure (COP) displacement assessed on force platform (BTS P-6000)
Functional Mobility | The outcome will assess at baseline and two weeks after the intervention. One month later that finished the intensive treatment subjects will re-evaluate.
  Evaluated by means of the Timed Up & Go Test (TUG)
Assessed by means of the Stroke-Specific Quality of Life Questionnaire (SSQOL) | The outcome will assess at baseline and two weeks after the intervention. One month later that finished the intensive treatment subjects will re-evaluate.
  The SSQOL questionnaire assesses the quality of life of stroke subject, and it contains 49 items with 12 domains (energy, family role, language, mobility, mood, personality, self-care, social role, reasoning, upper limb function, vision and work/productivity). There are three possible answers on the 5-point Likert scale.
  The SSOOL questionnaire score reports a minimum of 49 points and a maximum of 245 points. The lower values represent the more dependence and difficulty to perform tasks.
Muscular tone assessed by the Modified Ashworth Scale | The outcome will assess at baseline and two weeks after the intervention. One month later that finished the intensive treatment subjects will re-evaluate.
  Assessed by the Modified Ashworth Scale. This scale consists of 5 ordinal values ranging from 0 (no tonus increase) to 4 (stiffness).
Assessment of Sensorimotor Recovery After Stroke by Fugl-Meyer scale | The outcome will assess at baseline and two weeks after the intervention. One month later that finished the intensive treatment subjects will re-evaluate.
  Fugl-Meyer scale of lower limb impairment. The evaluation includes measurement of voluntary movement, velocity, coordination and reflex activity, through an ordinal scale applied to each item: 0- cannot be performed, 1- partially performed, and 2-performed completely. Participants were also classified according their LL motor impairment in severe (0 to19), moderate (20 to 28) or mild (> 29 points).
Serum levels of Brain-derived neurotrophic fator (BDNF). | The outcome will be assessed at baseline and 2 weeks after the intervention.
  The biomarker BDNF will be determined using the enzyme-linked immunosorbent assay (ELISA) method.
Serum levels of Insulin-like growth factor binding protein-3 (IGFBP-3) | The outcome will be assessed at baseline and 2 weeks after the intervention.
  The biomarker IGFBP-3 will be analyzed in the blood sample to evaluate the neuromuscular adaptations indirectly. Serum IGFBP-3 levels will be determined using the enzyme-linked immunosorbent assay (ELISA) method.
Serum levels of insulin-like growth factors 1 (IGF-1) | The outcome will be assessed at baseline and 2 weeks after the intervention.
  The IGF-1 will be analyzed in the blood sample to evaluate the neuromuscular adaptations indirectly. Serum IGF-1 levels will be determined using the enzyme-linked immunosorbent assay (ELISA) method.

CONTACTS AND LOCATIONS:
Overall Officials: Aline S Pagnussat, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] da Cunha MJ, Pinto C, Schifino GP, Sant'Anna Py I, Cimolin V, Pagnussat AS. Bicephalic Transcranial Direct-Current Stimulation Does Not Add Benefits to a Footdrop Stimulator for Improving Functional Mobility in People With Chronic Hemiparesis After Stroke: A Double-Blind, Randomized Controlled Trial. Phys Ther. 2022 Aug 4;102(8):pzac079. doi: 10.1093/ptj/pzac079. PMID 35689805